CLINICAL TRIAL: NCT06310395
Title: Analysis of the Acute Mesenteric Ischemia Management in a Single Institution Over 10 Years
Brief Title: Analysis of the Acute Mesenteric Ischemia in a Single Institution Over 10 Years
Acronym: AMI_HMAR
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Ana María González Castillo, Doctor, Hospital del Mar
Other Study IDs: AMI_H.MAR
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Acute Mesenteric Ischemia
Keywords: Mesenteric ischemia; Acute Mesenteric ischemia; Abdominal pain; Elderly; Complications; Mortality
MeSH Terms: conditions — Mesenteric Ischemia; Abdominal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute mesenteric ischemia (AMI) is a notorious disease with a high mortality, the diagnostic and management is truly multidisciplinary, but it is not the reality in many Hospitals.

The aim of this study is to analyse the results of the patients admitted with an AMI in Hospital de Mar.

DETAILED DESCRIPTION:
Acute mesenteric ischemia (AMI) is a notorious disease with a high mortality from 50 to 80%. Even though AMI is a relatively rare condition (1:1,000) the incidence rises exponentially with increasing age, in patients older than 75 years, the incidence of AMI has been reported higher than that of acute appendicitis. AMI patients benefit from early assessment in a surgical unit with capabilities to definitive management. The diagnosis and management of AMI are truly multidisciplinary, requiring high index of suspicion and awareness from emergency department physicians, preferably computed tomography angiography with precise interpretation.

The aim of this study is to analyse the results of the patients admitted with an AMI in Hospital de Mar from January 2014 to December 2023.

ELIGIBILITY:
Inclusion Criteria:

* Acute Mesenteric Ischemia

Exclusion Criteria:

* Chronic Mesenteric Ischemia
* Ischemic Colitis
* Bowel obstruction strangulation
* Inflamatory bowel necrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admited in Hospital del Mar from 2014 to 2023 with a diagnostic of AMI
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Mortality | 2014-2023
  To describe the mortality in patients with a diagnostic of AMI